CLINICAL TRIAL: NCT00563134
Title: A Prospective, Randomized, Double-blind, Placebo Controlled, Dose Ranging, Multi-Center Study of the Safety and Efficacy of Three Days Continuous Intravenous Infusion of GR270773 in the Treatment of Suspected or Confirmed Gram-negative Severe Sepsis in Adults
Brief Title: A Randomised Trial on the Saftely and Efficacy of GR270774 in the Treatment of Gram-negative Sepsis in Adult
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KW/FR/04-018; HARECCTR0500030
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Gram-Negative Bacterial Infections; Sepsis
Keywords: Suspected or confirmed severe Gram-negative sepsis
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Sepsis

INTERVENTIONS:
Drug: GR270774

SUMMARY:
Sepsis sometimes occurs in people who have a serious infection. It is caused by toxic substances (toxins) from bacteria and other germs entering your bloodstream. Most people with sepsis will recover with routine medical care before the illness gets more serious. However, in some people, sepsis does become more serious. This severe sepsis can cause damage to internal organs (such as your heart, lungs, kidneys, and liver) and can be life threatening. Special natural fats, (called 'lipoproteins') in our blood are thought to help protect us from the toxins produced by bacteria during sepsis. Levels of these lipoproteins are often low in people with sepsis and this may make it more difficult to recover from the disease. GR270773 is a new drug that has been developed to help the lipoproteins in protecting the body against toxins. GR270773 is made from purified fats and oils from the soyabean and does not contain cholesterol. This research study will test the safety (side effects) of GR270773 and whether or not it is effective in preventing complications in people with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or over.
* Subject has one of the following bacterial infections (as defined in Section 14.5) and a suspected or confirmed Gram-negative etiology:

  * Confirmed Gram-negative bacteremia (Gram-negative pathogen must be isolated from blood culture prior to study entry)
  * Intra-abdominal infection
  * Nosocomial pneumonia (Evidence of Gram-negative organism from histology or by direct stain of a respiratory specimen required prior to study entry)
  * Pyelonephritis
* Subject is receiving new parenteral antibacterial treatment for the suspected or confirmed Gram-negative infection believed to be responsible for this episode of sepsis. The subject must receive study drug within 36 hours of commencing treatment with this new antibacterial agent.

Note: Changes in antibiotic coverage made to treat the infection causing the current episode of sepsis or needed to treat a deteriorating subject in whom previous antibiotic coverage was deemed inadequate will be viewed as a new antibiotic.

* Subject has signs of new-onset severe sepsis as evidenced by at least ONE of the following hypoperfusion abnormalities OR organ failures caused by the current episode of sepsis. Subject must receive study medication within 12 hours from onset of the first sepsis-related hypoperfusion abnormality or organ failure:

  * Persistent oliguria (urine output <0.5 mL/kg/hr for at least two hours after adequate volume resuscitation (ie, >=2 L isotonic crystalloid or appropriate colloid to achieve the same effect)) Note: This criterion does not apply to subjects with chronic renal insufficiency/failure.
  * Metabolic acidosis (either a pH <=7.3 or a base deficit >5 mmol/L and a blood lactate level >2X the upper limit of normal)
  * Respiratory failure: PaO2/FiO2 <200
  * Coagulopathy: acute sepsis-related changes in either platelet count (<100,000 cells/mm3) or INR (>1.5)
  * Cardiovascular failure: sustained hypotension requiring vasopressor support (dopamine >5 µg/kg/min, epinephrine, norepinephrine, phenylephrine or vasopressin at any dose if used to increase blood pressure) for >1 hour in subjects in whom volume resuscitation is believed to be adequate (ie, subject has received >=2 L isotonic crystalloid or appropriate colloid to achieve the same effect) Note: Where a hypoperfusion abnormality/organ failure definition requires a condition to persist for a specified period of time, the organ failure is not considered to exist until the condition specified by the definition is met. The 12 hour window for start of study drug begins when the criteria for the organ failure/hypoperfusion are fulfilled. For organ failure/hypoperfusion abnormality defined in terms of a laboratory result (ie, metabolic acidosis, respiratory failure, and coagulopathy) the criteria for the organ failure/hypoperfusion are considered to be fulfilled at the time the laboratory sample was drawn. Otherwise, the 12 hour window begins at the time the organ failure definition criteria are fulfilled (ie, persistent oliguria and cardiovascular failure). Organ failures occurring subsequent to subject randomization but prior to initiation of study drug infusion do not constitute a secondary endpoint. These are treated as organ failures at study entry and should be documented as such in the relevant CRF pages. The occurrence of a subsequent organ failure does not redefine the start of the 12 hour window for start of study drug. This period is defined above to begin at the onset of the first sepsis-related organ failure qualifying the subject for study entry.
* Subject or their legally acceptable representative has provided written and dated informed consent to participate in the study.
* Subject, if female of childbearing potential or less than one year post menopausal (including those who are practicing birth control and those with tubal ligations), has a negative urine pregnancy test (measuring human chorionic gonadotropin(HCG) result prior to enrollment.

Exclusion Criteria:

* Subject is currently participating in or has participated in an investigational drug or medical device trial within 30 days or five half-lives, which ever is longer, prior to enrollment in this study.
* Subject is unlikely to remain in hospital for a minimum of three days (72 hours) following enrollment.
* Subject has neutropenia (e.g., subject recently receiving cytotoxic chemotherapy with absolute neutrophil count <500/µL or expected to decline to <500/µL in the next 3 days).
* Subject is known or believed to suffer from hereditary spherocytosis or S.E. Asian elliptocytosis.
* Subject has known active hemolytic disease; immune hemolytic anemias, hemoglobinopathies (sickle cell anemia and thalassemia major).
* Subject has a known bone marrow disorder of inadequate red cell production (eg, aplastic anemia, myelodysplasia).
* Subject is at increased risk of complications from GR270773-related hemolysis due to the inability to increase cardiac function sufficiently to meet the demands for oxygen delivery.
* Subject has a hemoglobin level at screening <9.0 g/dL (5.59 mmol/L). This hemoglobin assessment should be based on the most recent available data in the subject's medical record at the time of screening and is not used in the assessment of the hemoglobin stopping rule described in Section 6.2.2.
* Subject is currently being treated with Xigris (Drotrecogin alfa (activated)) or its use is considered imminent (ie, a decision to treat with Xigris has been made).
* Subject has a history of allergic reaction to eggs (or egg products), soybeans, Intralipid, or any component of GR270773.
* Subject has been designated as 'not full support', 'do not resuscitate' (DNR), or other equivalent status which prohibits the use of life supporting interventions (e.g., mechanical ventilation, dialysis/hemofiltration, or others) thereby limiting the treatment options available.

Note: Subjects with advanced directives prohibiting only chest compression (CPR) are eligible for the study.

* Subject has preexisting severe liver disease such as cirrhosis, primary biliary cirrhosis or known preexisting Child-Pugh class B or C liver dysfunction.
* Subject is moribund (a state in which death is perceived to be imminent) or has a life expectancy of less than 3 months due to an underlying disease.
* Subject is currently receiving one of the following prohibited concomitant medications; parenteral nutrition supplements containing lipid emulsions (eg, Intralipid), or systemic administration of amphotericin preparations (for example; amphotericin, liposomal amphotericin, or amphotericin B lipid complex).

Note: the use of topical amphotericin and oral amphotericin products are permitted and may be administered concomitantly with study drug at the discretion of the investigator.

* Subject is pregnant (positive urine pregnancy test at baseline) or lactating.
* Subject has previously been enrolled in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2005-10; Study Completion 2006-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days

SECONDARY OUTCOMES:
New onset organ failure | 28 days
Safety and tolerablity | 28 days
Long term mortality | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wai Chun Yip, Dr, Principal Investigator — Department of Surgery, Kwong Wah Hospital
Locations (1):
- Kwong Wah Hospital, Hong Kong, China